CLINICAL TRIAL: NCT00792558
Title: A Phase I Ascending Multiple-Dose Study of BMS-817378 in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: Ascending Multiple-Dose Study of BMS-817378 in Subjects With Advanced Cancers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA195-001
Record Dates: First submitted 2008-11-17; First posted 2008-11-18 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2009-01

CONDITIONS: Advanced Solid Tumors

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: BMS-817378

INTERVENTIONS:
Drug: BMS-817378 — Capsule, Oral, Dose escalation to a MTD from a starting dose of 25 mg, once daily, until disease progression/subject discontinuation

SUMMARY:
The purpose of this study is to find the maximum tolerated dose of BMS-817378 in subjects with advanced cancers

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of advanced non-hematologic malignancy. Dose expansion cohort restricted to subjects with advanced or metastatic gastroesophageal cancer, squamous cell cancers of the head and neck, and castration resistant prostate cancer
* ECOG status 0-1

Exclusion Criteria:

* WOCBP unwilling/unable to use acceptable contraception methods, and women pregnant or breast feeding
* Symptomatic brain metastasis
* Uncontrolled or significant cardiovascular disease
* History of thromboembolic events or bleeding diathesis in past 6 months
* Conditions requiring prophylactic anticoagulation or chronic anti-platelet therapy
* Serious non-healing wounds, ulcers or bone fractures in past 3 months
* Hemorrhage or bleeding event >= CTCAE grade 3 in past 4 weeks
* Proteinuria >= 2+ on dipstick or >= 1gm/24 hours
* Concurrent chemotherapy, hormonal therapy, immunotherapy, radiation therapy or therapy with any other investigational product
* Concurrent herbal, alternative, food supplements, or strong CYP 3A4 inhibitors or inducers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2010-11 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
To establish the MTD of BMS-817378 when administered orally on a daily schedule in subjects with advanced cancers | Within the first 21 days after first dose of BMS-817378

SECONDARY OUTCOMES:
Assess safety and tolerability of multiple doses of BMS-817378 administered orally on a once daily schedule in subjects with advanced or metastatic solid tumors | All time points while subject is on study
Assess the safety and tolerability of co-administration of a CYP substrate cocktail and BMS-817378 given at or below the MTD (dose expansion cohort) | Day 22 +/-2
Characterize the pharmacokinetics of BMS-817378 and its active moiety, BMS-794833 | Days 1 and 15
Assess the effects of BMS-817378 and BMS-794833 on blood pressure, heart rate, ECG intervals, and left ventricular ejection fraction | All time points while subject is on study
Describe preliminary evidence for anti-tumor activity of BMS-817378 | Every 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- Australia (2):
  - Local Institution, Adelaide, South Australia
  - Local Institution, Nedlands, Western Australia
- Local Institution, Singapore, Singapore